CLINICAL TRIAL: NCT01362660
Title: A Protocol to Monitor the Neurological Development of Infants With Exposure In-utero From Birth to Aged 15 Months in Tanezumab Clinical Studies at Investigational Sites Overseen by Schulman and Associates Institutional Review Board
Brief Title: A Study to Evaluate Infants With Potential Exposure to Tanezumab Before Birth
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4091055; NEONATAL MONITORING
Record Dates: First submitted 2011-05-24; First posted 2011-05-30 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Infant Developmental Assessment
Keywords: post-natal monitoring; exposure in utero

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infants with potential exposure in utero
  Interventions: Other: Unintentional exposure in utero

INTERVENTIONS:
Other: Unintentional exposure in utero — This study will examine post-natal neurologic and cognitive development of infants who may have been exposed to tanezumab or comparator in-utero during the tanezumab clinical program (whether the exposure is through maternal or paternal participation in a tanezumab clinical study).

SUMMARY:
This study will examine post-natal neurologic and cognitive development of infants who may have been exposed to tanezumab or comparator in-utero during the tanezumab clinical program (whether the exposure is through maternal or paternal participation in a tanezumab clinical study).

DETAILED DESCRIPTION:
This study will enroll infants with potential tanezumab exposure in utero at sites overseen by Schulman and Associates IRB This study will attempt to enroll all infants who qualify.

ELIGIBILITY:
Inclusion Criteria:

Subject is an infant born to a mother who was exposed to study drug on a tanezumab clinical study through direct maternal exposure; or is an infant born to a mother who is a partner of a male patient who was exposed to study drug in a tanezumab clinical study prior to or around the time of conception and/or is exposed during his partner's pregnancy.

Exclusion Criteria:

There are no exclusion criteria for this study

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with potential exposure in utero through their parents partcipation in a tanezumab clinical study
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Bayley Infant Neurodevelopmental Screener | 0-2 Months
Bayley Infant Neurodevelopmental Screener | 8 months
Bayley Infant Neurodevelopmental Screener | 15 months
Receptive-Expressive Emergent Language Test | 0-2 Months
Receptive-Expressive Emergent Language Test | 8 months
Receptive-Expressive Emergent Language Test | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Wildomar, California
  - Pfizer Investigational Site, Cutler Bay, Florida
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091055&StudyName=A%20Study%20to%20Evaluate%20Infants%20with%20Potential%20Exposure%20to%20Tanezumab%20Before%20Birth%20